CLINICAL TRIAL: NCT03973697
Title: A Phase II, Randomized Trial to Evaluate the Optimal Dosing of Fecal Microbiota Transplantation Using the Penn Microbiome Therapy Products for Recurrent Clostridium Difficile Infection
Brief Title: Penn Microbiome Therapy for Recurrent Clostridium Difficile Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 832963
Record Dates: First submitted 2019-04-17; First posted 2019-06-04 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Intervention Model Description: Randomized, open label, comparative
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single dose of PMT (Experimental)
  Interventions: Drug: Penn Microbiome Therapy - 001; Drug: Penn Microbiome Therapy - 002; Drug: Penn Microbiome Therapy - 003
- Two doses of PMT (Experimental): Administered within 24 hours
  Interventions: Drug: Penn Microbiome Therapy - 001; Drug: Penn Microbiome Therapy - 002; Drug: Penn Microbiome Therapy - 003

INTERVENTIONS:
Drug: Penn Microbiome Therapy - 001 — Fecal Microbiota for Transplant, enema product
  Other Names: PMT-001
Drug: Penn Microbiome Therapy - 002 — Fecal Microbiota for Transplant, suspension product
  Other Names: PMT-002
Drug: Penn Microbiome Therapy - 003 — Fecal Microbiota for Transplant, capsule product
  Other Names: PMT-003

SUMMARY:
This is a randomized, open label, comparative, Phase II study to determine which dose of fecal microbiota transplant using Penn Microbiome Therapy (PMT) products is most effective in treating and preventing recurrence of Clostridium difficile infection (C diff).

ELIGIBILITY:
Inclusion Criteria:

1. Second or greater episode of CDI (first or greater recurrence) within 12 months, with symptoms including bowel movement altered in frequency or consistency from baseline.
2. Stool positive for C. difficile toxin by EIA or toxin gene by NAAT within 60 days of enrollment.
3. At least one additional prior positive stool test for C. difficile within the prior 12 months (EIA or NAAT as above).
4. Age ≥ 18 years.
5. Minimum of 72 hours of receipt of standard-of-care (vancomycin or fidaxomicin) antibiotic treatment for R-CDI prior to intervention.

Exclusion Criteria:

1. Evidence of colon/small bowel perforation at the time of study screening
2. Goals of care are directed to comfort rather than curative measures.
3. Moderate (ANC < 1000 cells/uL) or severe (ANC < 500 cells/uL) neutropenia.
4. Known food allergy that could lead to anaphylaxis.
5. Pregnancy

   a. For subjects of childbearing potential (ages 18 to 55), the subject must have a negative urine pregnancy test within 48 hours of consent and no more than 48 hours prior to first product administration
6. Meeting criteria for severe, severe-complicated/fulminant CDI within 24 hours of planned trial enrollment. We define severe or severe-complicated/fulminant CDI as any one of the following: (1) leukocytosis with peripheral WBC ≥ 15,000 cells/mL; (2) hypotension with systolic blood pressure sustained < 90mmHg for three or more hours or requiring pressors; (3) provider documentation of ileus or radiologic evidence of bowel dilation or megacolon; (4) acute kidney injury with increase in baseline serum creatinine level by ≥50% or new dialysis initiation; (5) serum lactate > 2.2 mmol/L; or (6) ≥ 3 systemic inflammatory response syndrome (SIRS) criteria (which include heart rate > 90 beats per minute, respiratory rate > 20 breaths per minute or PaCO2 < 32 mmHg, temperature >38ºC or <36ºC, WBC > 12,000 cells/uL, <4,000 cells/uL, or >10% immature (band) forms).
7. Receipt of FMT or enrollment in a clinical trial for FMT within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebbing Lautenbach, MD, MPH, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the Univeristy of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Dose of PMT | Two Doses of PMT
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose of PMT | Two Doses of PMT | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Resolution of Symptoms After Treatment With One of the PMT Suite of Products or Control.
Description: Clinical resolution will be compared by determining the proportion of subjects with clinical resolution of diarrhea without recurrence in subjects with R-CDI at 8 weeks (56 days) following FMT. Clinical resolution will be defined as follows:
  * ≤ 4 stools per calendar day for the prior two days with no stool of Bristol stool scale type 7
  * No additional stool tests with a positive EIA for C. difficile toxin since study enrollment
  * No additional prescription or use of anti-CDI antibiotics (unless given for prophylaxis) since study enrollment
  * No need for an additional
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PMT | Two Doses of PMT
Number analyzed (Participants) | 5 | 4
Participants | 1 | 2

2. Secondary Outcome: All-cause Mortality at 30-days Following Last FMT
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PMT | Two Doses of PMT
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

3. Secondary Outcome: All-cause Mortality at 60-days Following Last FMT
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PMT | Two Doses of PMT
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

4. Secondary Outcome: Colectomy or Diverting Ileostomy Within 30 Days After Last FMT
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PMT | Two Doses of PMT
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

5. Secondary Outcome: Cumulative Days of Hospitalization From Enrollment Until 30 Days After FMT
Time Frame: 30 days
Measure: Median (Full Range); unit: days
Arm/Group | Single Dose of PMT | Two Doses of PMT
Number analyzed (Participants) | 5 | 4
days | 10 [5 to 16] | 1 [1 to 1.5]

6. Secondary Outcome: Cumulative Days in Intensive Care Unit From Enrollment Until 30 Days After Last FMT
Time Frame: 30 Days
Measure: Median (Full Range); unit: days
Arm/Group | Single Dose of PMT | Two Doses of PMT
Number analyzed (Participants) | 5 | 4
days | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Bacteremia From Enrollment Until 30 Days After Last FMT
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PMT | Two Doses of PMT
Number analyzed (Participants) | 5 | 4
Participants | 1 | 0

8. Secondary Outcome: Hospital Admission Within 60 Days of Discharge From Index Hospitalization
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose of PMT | Two Doses of PMT
Number analyzed (Participants) | 5 | 4
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Dose of PMT | Two Doses of PMT
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/5 | 3/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose of PMT (N=5) | Two Doses of PMT (N=4)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diahrrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders-other (Gastrointestinal disorders) | 1 (1) | 0 (0) — IBS/Crohn's
Gastrointestinal disorders-other (Gastrointestinal disorders) | 0 (0) | 1 (1) — Venrtal hernia
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Surgical and medical procedures-other (Surgical and medical procedures) | 0 (0) | 1 (1) — right total hip arthroplasty
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose of PMT (N=5) | Two Doses of PMT (N=4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders-other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Leukopenia
Blood and lymphatic system disorders-other (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Thrombocytopenia
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Ascites (Gastrointestinal disorders) | 2 (3) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (4)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 2 (9)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders-other (Gastrointestinal disorders) | 0 (0) | 1 (1) — increased frequency of bowel movement
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Investigations-Other (Investigations) | 1 (1) | 0 (0) — Bacteremia
Investigations-other (Investigations) | 0 (0) | 1 (1) — HIV viral load change
Lipase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — squamous cell carcinoma
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 (1) | 1 (1) — decreased urinary frequency
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Otitis media (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
skin and subcutaneous tissues disorders-other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — oral lesion
skin and subcutaneous tissue disorders-other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Peri-rectal erythema
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03973697/Prot_SAP_000.pdf